CLINICAL TRIAL: NCT05357248
Title: Nutritional Cognitive Behavioral Therapy Feasibility Study in NAFLD and NASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Better Therapeutics (Industry)
Collaborators: Arizona Liver Health (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT-NCBT-00x
Record Dates: First submitted 2022-04-27; First posted 2022-05-02 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Non-alcoholic Steatohepatitis; Non-Alcoholic Fatty Liver Disease; Non-alcoholic Fatty Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: This single arm study of 20 patients is to evaluate the feasibility of using BT-NCBT-00x in the treatment of NAFLD and NASH
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Intervention- BT-NCBT-00x (Experimental): The treatment, BT-NCBT-00x, consists of a software as a medical device developed by the study Sponsor, Better Therapeutics. It delivers treatment to participants with cardiometabolic disease, using behavioral therapy that targets individual behaviors related to improving dietary quality and physical activity. BT-NCBT-00x is accessed via the participants' smartphone after downloading from the phone's corresponding app store.
  Participants will receive behavioral support by the Better Therapeutics patient services team in the form of phone calls as necessary or requested by the patient
  Interventions: Device: BT-NCBT-00X

INTERVENTIONS:
Device: BT-NCBT-00X — the intervention group will consist of 20 patients to receive the BT-NCBT-00X treatment for 90 days. They will receive a baseline MRI-PDFF, Fibroscan and have the tests repeated at 90 days.

SUMMARY:
This single arm interventional cohort study is designed to explore the feasibility of using BT-NCBT-00x to improve liver fat, inflammation, and stiffness in patients diagnosed with NAFLD or NASH over a 3 month intervention.

DETAILED DESCRIPTION:
The treatment, BT-NCBT-00x, consists of a software as a medical device developed by the study Sponsor, Better Therapeutics. It delivers treatment to participants with cardiometabolic disease, using behavioral therapy that targets individual behaviors related to improving dietary quality and physical activity. The study evaluates the use of this behavioral therapy and its effect on clinical measures such as percent liver fat as measured by MRI-PDFF, and Fibroscan Controlled Attenuation Parameter score, liver stiffness as measured by Fibroscan Vibration Controlled Transient Elastography in kPA, body weight and ALT. Participants in this feasibility study will have access to the treatment for 3- months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NAFLD or NASH
* At least 2 doses of the COVID-19 Vaccine, per self report
* Possession of a smartphone capable of running the Bt_NCBT-00x application
* BMI >/= 30 at the screening visit
* Fibroscan CAP >300 dB/m collected at screening visit
* Completion of baseline MRI-PDFF
* Understand written and spoken english

Exclusion Criteria:

* Inability to read and understand english
* unstable or life-threatening medical illness
* weight loss of greater than 10lbs within the last 90 days
* pregnant or planning to become pregnant women
* concurrent enrollment in any other interventional clinical trial
* presumed or confirmed COVID-19 diagnosis within 30 days prior to study enrollment
* change in medication regimen of hormonal contraceptives, anti-hyperglycemic medications, mental or emotional disorder medications, corticosteroids, thyroid hormones, Tamoxifen or Methotrexate within 90 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
change in percent liver fat | 90 days
  Mean change in percent liver fat from baseline to end of treatment in participants with baseline PDFF ≥ 10%, as measured by MRI-PDFF.

SECONDARY OUTCOMES:
Change in Liver Fat- all participants | 90 days
  Mean change in liver fat from baseline to end of treatment in all participants, as measured by MRI-PDFF
Reduction in Percent Liver fat | 90 days
  Percent of participants who achieve ≥ 30% change in PDFF from baseline to end of treatment

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Arizona Liver Health, Chandler, Arizona
  - Arizona Liver Health, Peoria, Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alkhouri N, Edwards K, Berman M, Finn H, Escandon R, Lupinacci P, Guthrie N, Coste A, Topete J, Noureddin M. A Novel Prescription Digital Therapeutic Option for the Treatment of Metabolic Dysfunction-Associated Steatotic Liver Disease. Gastro Hep Adv. 2023 Oct 1;3(1):9-16. doi: 10.1016/j.gastha.2023.08.019. eCollection 2024. PMID 39132187